CLINICAL TRIAL: NCT00734422
Title: Facilitation of Fear Extinction With Yohimbine Hydrochloride in Phobic Participants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KP-2007-226
Record Dates: First submitted 2008-08-11; First posted 2008-08-14 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Phobic Disorders
Keywords: Phobic Disorders (Fear of Flying); Virtual Reality Exposure Therapy; Fear extinction; Yohimbine
MeSH Terms: conditions — Phobic Disorders; Aerophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRET with yohimbine (Experimental): Virtual Reality Exposure Therapy will be combined with the administration of yohimbine hydrochloride
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- VRET with placebo (Placebo Comparator): Virtual Reality Exposure Therapy will be combined with an inactive placebo pill (Albochin).
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Standard virtual reality exposure therapy for fear of flying will be combined with the administration of either yohimbine hydrochloride or an inactive placebo pill.

SUMMARY:
Procedurally Virtual reality exposure therapy (VRET) is quite similar to models of extinction of conditioned fears. Recent advances in animal research have identified pharmacological agents that appear to both accelerate and consolidate extinction learning. One of these cognitive enhancers is Yohimbine. An interesting finding in animal literature is that the administration of Yohimbine during extinction trials accelerates fear reduction and may convert ineffective exposures in to successful ones. It is thought that the mechanism of enhanced emotional memory is through elevated norepinephrine in the prefrontal cortex. Therefore, we propose to extend these studies by combining VRET with Yohimbine. In this pilot study with a between groups design 20 participants with a fear of flying will be treated with VRET plus Yohimbine or VRET plus placebo. This between groups design was chosen to further characterize the differential within and between trial extinction. Outcome will be measured by self-report, behavioral, and psychophysiological assessments at pre- and post-treatment. In addition, we will examine extinction parameters during exposures.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of specific phobia (fear of flying).
* Between the ages of 18-65
* Sufficient fluency in Dutch to complete treatment and research protocol

Exclusion Criteria:

* Presence of medical condition, assessed by self-report questionnaires at the intake (i.e., pregnancy, seizure disorder, respiratory disorder, cardiovascular disease, pacemaker, hypertension).
* Resting blood pressure higher than 140 (systolic) or 105 (diastolic)
* Unstable psychotropic medication.
* Current use of tranquilizers (Benzodiazepines)
* Psychosis
* Depression with suicidal ideation
* Dementia or other severe cognitive impairment
* Substance dependence
* Bipolar disorder
* Borderline personality disorder
* Anti-social personality disorder
* Current use of beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Flight Anxiety Situations Questionnaire (self-report); Flight Anxiety Modality Questionnaire (self-report) | Assessed at pre- and post-treatment and 9-12 months follow-up

SECONDARY OUTCOMES:
Severity of Anxiety Symptoms (Beck Anxiety Inventory) Anxiety Sensitivity (Anxiety Sensitivity Inventory) | Assessed at pre- and post-treatment and 9-12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul MG Emmelkamp, Professor, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, Netherlands